CLINICAL TRIAL: NCT07158983
Title: Evaluation of a Child Health Care Program for Early Identification of Family Violence
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Forte: Swedish research council for health, working life and welfare (Unknown)
Responsible Party: Principal Investigator, Lene Lindberg, Professor, Karolinska Institutet
Other Study IDs: FRIDa
Record Dates: First submitted 2025-08-20; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Identification of Family Violence
Keywords: Family violence; Parental support; Identification; Screening; Primary health care; Evaluation
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents: Parents of children enrolled in child health services
  Interventions: Other: Registry review
- Nurses: Nurses working within child health services
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Registry review — The study is set within a project to evaluate a program for identification of family violence. The study uses mixed methods including registry review of parents to evaluate the effect of the program.
  Groups: Parents
Other: Interviews — The study is set within a project to evaluate a program for identification of family violence. The study uses mixed methods including interviews with nurses to evaluate the effect of the program.
  Groups: Nurses

SUMMARY:
The aim of this mixed methods study is to gain knowledge about how a program for identification of family violence works within child health services. The main research questions are:

* To what extent are questions about family violence asked to mothers and fathers visiting the child health services in the Region of Stockholm?
* How can area level socioeconomic factors affect whether parents are asked questions about family violence in the child health services?
* How do child health nurses experience asking parents about family violence?What challenges and opportunities do they meet when they identify family violence?

DETAILED DESCRIPTION:
Being exposed to family violence (FV) as a child is associated with an increased risk of negative impact on development and health both in the short and long term. Research shows that FV occurs in all cultures and in all social classes. However, there is an increased risk of FV in areas with a higher degree of social vulnerability. For children, FV means being directly exposed to psychological, physical, sexual violence or neglect. It can also mean experiencing violence between adults in the home, which leads to the same negative consequences for the child. Parents with current or previous experiences with FV have an increased risk of difficulties in parenting skills, which in turn can affect the child negatively.

In Sweden, almost all children 0-5 years old are enrolled in the child health services (CHS). As part of the CHS-program, all parents are offered an individual visit within the first six months of their child's life to address parenting topics and parental mental health. Questions about FV are asked during that individual visit. The CHS thus has a unique opportunity to detect FV in the family at an early stage in the child's life.

This mixed methods study evaluates how a program for identification of family violence works within child health services. The quantitative part is a registry based observational study to investigate the extent to which both mothers and fathers are given the opportunity to respond to questions about FV within CHS in the Stockholm region. Furthermore, it examines whether there is an association between being asked about exposure to violence and the socioeconomic status of the catchment areas of CHS centers. The qualitative data consist of interviews with child health nurses.

De-identified medical record data regarding questions about family violence addressed to the child's parents will be collected from approximately 90,000 child records at the CHS centers. Included CHS centers are located in areas with different socioeconomic status. Data cover the period 240630-250630. Background data on the organizational conditions (number of employees, training to identify FV) of the included CHS centers are also obtained. The results are also measured based on the clinic's sociodemographic, according to the Care Need Index (CNI). The data enables comparisons between different CHS centers, and the interviews contributes to an in-depth analysis of the study's results based on varying contextual factors that may assist or hinder the identification of FV.

ELIGIBILITY:
Inclusion Criteria:

* Parents to children enrolled in the CHS
* Child health nurse working at one of the included CHS centers

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population are parents to children enrolled in CHS in the Stockholm region and nurses working in CHS in the Stockholm region
Sampling Method: Non-Probability Sample
Enrollment: 90000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Parents being asked about family violence according to patient records | 1 year
  Mothers and fathers who have been asked about family violence at the child health services according to the child's patient record (yes/no)
Nurses experiences of opportunities and challenges in the work around family violence identified through qualitative assessments | Time since the program was implemented, between three and five years
  Nurses are asked about opportunities and challenges to pose questions about family violence. They are invited to share their experiences about identifying family violence and offering support.

SECONDARY OUTCOMES:
Identification of family violence documented in patient records | 1 year
  Identification of family violence among parents and children enrolled at the CHS (yes/no)
Reports to the social services documented in patient records | 1 year
  Reports to the social services filed by nurses due to identified family violence documented in patient records

CONTACTS AND LOCATIONS:
Overall Officials: Lene Lindberg, Professor, Principal Investigator — Karolinska Institutet: Department of Global Public Health
Locations (1):
- Region Stockholm, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
IDP are not avialable due to the ethical approval. Access to data requires ethical approval and could then be provided upon request.